CLINICAL TRIAL: NCT00507533
Title: Early Application of CPAP in Hematologic Neutropenic Patients Avoid Acute Respiratory Failure
Brief Title: Early Application of CPAP in Hematologic
Acronym: HEMOCPAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPAP-2-H
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Hematologic Disease
Keywords: CPAP; Hematologic; Neutropenic; ARF
MeSH Terms: conditions — Hematologic Diseases | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Continuous positive airway pressure

SUMMARY:
The purpose of this study is to evaluate the use of CPAP in the prevention of acute respiratory failure in neutropenic ( or hematologic malignancy ) patients .CPAP applied preventively in hematological patients with high risk of ARF may reduce:need for intubations and mechanical ventilation, incidence of pneumonia and sepsis,mortality,length of ICU and hospital stay

DETAILED DESCRIPTION:
Immunocompromised patients with a hematological malignancy that requiring admission in intensive care unit (ICU) and subsequently mechanical ventilation for respiratory failure was estimated between 20- 50 per cent of all admitted in hospital.

The survival rate of this patients that requiring mechanical ventilation is very poor.

In many cases the immunodepression with a great improvement in severe complication as infections , pneumonia, sepsis , is the consequence of our therapy ( chemotherapy , bone marrow transplantation and stem cell transplantation ) .

Pneumonia is very common cause of mechanical ventilation in about 45-74 per cent of the all patient with acute respiratory failure (ARF) .

The trial was designed to enroll 40 patients in two groups to demonstrate reduction from 50% to 10 % of the need of mechanical ventilation , with a type I risk of error of 5% and a power of 80 %.

Patients were randomized to be treated for four days Venturi mask at a FiO2 of 0.4 (control) or with oxygen at a FiO2 of 0.4 plus a CPAP of 10 cm H2O (CPAP). At the end of the 4-days period, patients passed a screening test breathing ambient air. Patients returned to the assigned treatment if SaO2 less than 95% a.a or respiratory rate more than 25 bpm.CPAP was generated using a flow generator with an adjustable inspiratory oxygen fraction set to deliver a flow of up to 140 liters per minute (Whisperflow, Caradyne, Ireland) and a spring-loaded expiratory pressure valve (Vital Signs Inc, Totoma NJ) and applied using a latex-free polyvinyl chloride transparent helmet (CaStar, Starmed, Italy) (15); all centers measured the inspiratory oxygen fraction using an oxygen analyzer (Oxicheck, Caradyne, Ireland) through the Venturi mask or the helmet.

ELIGIBILITY:
Inclusion Criteria:

* Neutropenic hematological patients ( less than 1000 leukocytes /mm3 ) .
* SaO2 less than 95% ( a.a.) ,
* Respiratory rate (RR ) more than 25 breaths/minute .

Exclusion Criteria:

* NYHA class II- III- IV or unstable angina or MI
* Valvular heart disease or cardiac surgery ( previous 3 months)
* Implanted cardiac pacemaker
* BMI less than 40
* History of dilated cardiomyopathy or CPE
* Severe COPD ( oxygen therapy , recent exacerbation, hypoxemic-hypercapnic to resting , FEV1 < 50 %)
* Diagnosis of sleep or neuromuscular disorders.
* Claustrophobia .
* Mechanical ventilation criteria:

  * Severe hypoxemia (arterial oxygen saturation < 80 % with maximal FiO2 )
  * Ph < 7.3 with a PaCO2 > 50 mmHg
  * Signs of patient distress with accessory muscle recruitment and paradoxal abdomen movement
  * RR > 35 breaths/minute .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
mechanical ventilation and intubation

SECONDARY OUTCOMES:
Pneumonia , sepsis , ICU LOS , Hospital LOS , Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Squadrone Vincenzo, MD, Principal Investigator
Locations (1):
- Università degli Studi Torino, Turin, Piedmont, Italy